CLINICAL TRIAL: NCT03280914
Title: Epidemiology and Intervention of Obstructive Sleep Apnea Based on Community: a Real World Study
Brief Title: Epidemiology and Intervention of Obstructive Sleep Apnea Based on Community
Status: Completed | Type: Observational
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: GDREC2016275H(R1)
Record Dates: First submitted 2017-08-14; First posted 2017-09-13 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2018-06

CONDITIONS: Sleep Apnea, Obstructive; Hypertension; Obesity; Diabetes; Hyperdiploid; Fatigue Syndrome, Chronic; Insomnia Chronic; Quality of Life; Economic Problems; Compliance, Patient; Health Impairment
Keywords: obstructive sleep apnea; real world; community
MeSH Terms: conditions — Sleep Apnea, Obstructive; Hypertension; Obesity; Diabetes Mellitus; Fatigue Syndrome, Chronic; Sleep Initiation and Maintenance Disorders; Patient Compliance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum lipid, glucose.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CPAP group: Automatic Continuous Positive Airway Pressure treatment and usual care
  Interventions: Device: Auto-CPAP
- Usual care group: Usual care without Continuous Positive Airway Pressure treatment

INTERVENTIONS:
Device: Auto-CPAP — Automatic Continuous Positive Airway Pressure treatment is the first-line treatment of obstructive sleep apnea
  Groups: CPAP group

SUMMARY:
This observational study in a real-world community was designed to perform epidemiological investigation and assess effect of CPAP intervention of obstructive sleep apnea.

DETAILED DESCRIPTION:
Patients with obstructive sleep apnea receiving CPAP or not would be observed in years. Primarily Impact of CPAP on health assessment andx control rate of hypertension would evaluated.

ELIGIBILITY:
Inclusion Criteria:

1) AHI >= 5 events/h

Exclusion Criteria:

1. Any condition which in the opinion of researched makes the eligible participants unsuitable for this study, such as severe COPD, heart failure in NYHA class III to IV, and others
2. Any condition potentially precluding follow-up visits, such as sereve insomnia, cognitive behavioral disorder, and others
3. Patients receiving CPAP treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients would be recruited from Community of Huanghua Road.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Health assessment | From 1st Aug 2017 to 31st Dec 2020
  Health assessment would be performed by 36-Item Short-Form Health Survey.
Sleep quality | From 1st Aug 2017 to 31st Dec 2020
  Sleep quality would be performed by Pittsburgh Sleep Quality Index.
Psychological assessment | From 1st Aug 2017 to 31st Dec 2020
  Psychological assessment would be performed by Hospital Anxiety and Depression Scale.
Control rate of hypertension | From 1st Aug 2017 to 31st Dec 2020

SECONDARY OUTCOMES:
Incidence of chronic diseases | From 1st Aug 2017 to 31st Dec 2025
  Chronic diseases include hypertension, coronary heart disease, stroke and diabetes.
Death from all-cause | From 1st Aug 2017 to 31st Dec 2025
Medical cost | From 1st Aug 2017 to 31st Dec 2025
  Medical fee, annually time of outpatient visit and hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Qiong Ou, M.D., Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Community of Huanghua Road, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No
Previous research plan submitted to the Ethics Committee has stated the participant information not be shared.